CLINICAL TRIAL: NCT02299323
Title: Circumferential Lumbar Spinal Fusion for Treatment of Degenerative Disc Disease: A Prospective, Non-Randomized Clinical Study
Brief Title: INDEPENDENCE Spacer for Lumbar Fusion
Status: Completed | Type: Observational
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RGC11-010-001-PL_C
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: INDEPENDENCE — Lumbar Integrated plate and spacer, with percutaneous screws and rods.

SUMMARY:
The primary objective of this study is to evaluate radiographic outcomes, intra-operative parameters, clinical outcomes, and patient satisfaction following circumferential fusion using the INDEPENDENCE® integrated plate and spacer with REVOLVE® Stabilization System for the treatment of severe low back pain due to lumbar disc degeneration unresponsive to 6 months of non-operative treatment.

DETAILED DESCRIPTION:
A total of thirty subjects will be enrolled at Scott & White Healthcare. The INDEPENDENCE spacer will be filled with autogenous bone graft material. The devices subject to this Agreement have received 510(k) clearance from the FDA for the indications specified in this Agreement.

Patients will be followed for 2 years with evaluations at the following time intervals: preoperatively (within 2 months of surgery) and postoperatively at 6 weeks, 3 months, 6 months, 12 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* • Objective evidence of degenerative disc disease at 1 or 2 level(s) between L2 and S1 with degeneration confirmed by patient history and radiographic examination

  * Experience pain, functional deficit and/or neurological deficit for a minimum of six months
  * Unresponsiveness to documented non-surgical treatment modalities for a minimum of six months and/or presentation with progressive symptoms of nerve root or spinal cord compression prior to enrollment
  * At least 18 years of age and maximum 65 years of age
  * Ability to provide Informed Consent for study participation and to return for all follow-up visits

Exclusion Criteria:

* • Presence of systemic or localized infection at the site of surgery

  * More than 2 levels to be instrumented
  * Previous fusion attempt at the involved level(s)
  * More than three previous open, posterior, lumbar spinal surgical procedures at the involved level(s)
  * Trauma at the level(s) to be fused
  * More than grade 1 spondylolisthesis
  * Previous documentation of osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated
  * Diagnosis of a condition or requires postoperative medication(s), which may interfere with bony/soft tissue healing
  * Presence of a disease entity or condition which totally precludes possibility of bony fusion (e.g. metastatic cancer, HIV, long term use of steroids, etc.)
  * Immunosuppressive disorder
  * Pregnant or interested in becoming pregnant during the duration of the study
  * History of substance abuse (drugs or alcohol)
  * Any known allergy to a metal alloy
  * Mentally incompetent or prisoner
  * Currently a participant in another study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between ages 18 and 65 withsevere low back pain due to lumbar disc degeneration unresponsive to 6 months of non-operative treatm
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Radiographic fusion evaluation | 2 years
  Anterior Posterior / Lateral, Flexion-Extension X-rays at every timepoint will be evaluated for signs of fusion, pseudoarthrosis and implant subsidence or migration

SECONDARY OUTCOMES:
Patient Self- Assessment for pain scores | 2 years
  VAS questionnaires to be completed at every follow-up timepoint
Patient Satisfaction | 2 years
  Questionnaire to be completed at every follow-up timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chaput, MD, Principal Investigator — Scott & White Healthcare
Locations (1):
- Scott & White Healthcare, Temple, Texas, United States